CLINICAL TRIAL: NCT01564186
Title: Characterization of Cardiac Hemodynamics by Pressure-Volume Loop Analysis During MultiPoint Pacing
Brief Title: Characterization of Cardiac Hemodynamics During MultiSite Pacing
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 643
Record Dates: First submitted 2012-03-24; First posted 2012-03-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MulitPoint Pacing
- BiV Conventional

SUMMARY:
The purpose of this study is to evaluate the effects of MultiPoint Pacing (MPP) on cardiac hemodynamics assessed by pressure-volume loop during MPP at implant. NYHA functional class assessment and echocardiographic measurements are performed at 3 months and 12 months post-implant to characterize long-term effect of MPP.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to undergo implant of a St Jude Medical CRT-D system with approved standard indication by ESC/EHRA Guidelines
* Be in sinus rhythm at the time of enrollment
* Have the ability to provide informed consent for study participation and be willing and able to comply with the Clinical Investigation Plan (CIP) described evaluations and follow-up schedule

Exclusion Criteria:

* Exhibit Cheyne-Stokes respiration
* Have persistent or permanent atrial fibrillation
* Have complete heart block
* Be in NYHA IV functional class
* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures in the following 7 months
* Have had a recent CVA or TIA within 3 months prior to enrollment
* Have had intravenous inotropic support in the last 30 days
* Be less than 18 years of age
* Be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for standard CRT-D therapy.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Within-patient differences in PV loop-based hemodynamic parameters (dP/dtMax, stroke work, stroke volume, ejection fraction) | At implant

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Italy

REFERENCES:
- [Derived] Pappone C, Calovic Z, Vicedomini G, Cuko A, McSpadden LC, Ryu K, Jordan CD, Romano E, Baldi M, Saviano M, Pappone A, Vitale R, Catalano C, Ciaccio C, Giannelli L, Ionescu B, Petretta A, Fragakis N, Fundaliotis A, Tavazzi L, Santinelli V. Improving cardiac resynchronization therapy response with multipoint left ventricular pacing: Twelve-month follow-up study. Heart Rhythm. 2015 Jun;12(6):1250-8. doi: 10.1016/j.hrthm.2015.02.008. Epub 2015 Feb 9. PMID 25678057
- [Derived] Pappone C, Calovic Z, Vicedomini G, Cuko A, McSpadden LC, Ryu K, Romano E, Baldi M, Saviano M, Pappone A, Ciaccio C, Giannelli L, Ionescu B, Petretta A, Vitale R, Fundaliotis A, Tavazzi L, Santinelli V. Multipoint left ventricular pacing in a single coronary sinus branch improves mid-term echocardiographic and clinical response to cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2015 Jan;26(1):58-63. doi: 10.1111/jce.12513. Epub 2014 Sep 19. PMID 25109276